CLINICAL TRIAL: NCT07292051
Title: Effect of Blood Flow Restriction Technique on Postpartum Pelvic Girdle Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nour Abdelaty Attia El-desouky, Physical Therapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-813
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): Group (A) will receive a core stability exercise program.
  Interventions: Other: Core Stability Exercise
- Group (B) (Experimental): Group (B) will receive core stability exercise program with blood flow restriction technique.
  Interventions: Other: Core Stability Exercise; Other: Blood Flow Restriction Technique

INTERVENTIONS:
Other: Core Stability Exercise — Patients will receive specific core stabilizing exercises, focusing on Pelvic floor muscles ,Gluteus maximus, Gluteus Medius, specific abdominal muscles , the lumbar multifidus, and Erector spinae.
Other: Blood Flow Restriction Technique — Patients will receive the same core stability exercise added to Blood Flow Restriction Technique
  Arms: Group (B)

SUMMARY:
Purpose of the study :

The purpose of the current study is investigating the effect of Blood Flow Restriction Training technique on postpartum pelvic girdle pain.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. To fulfill its purpose, we have two groups; control group (A) and experimental group (B) are two matched postpartum pelvic girdle pain groups. While group (A) will receive a core stability exercise program, group (B) will receive core stability exercise program with blood flow restriction technique.

The primary outcome measure will be pelvic girdle pain intensity, while the secondary outcomes will include pelvic girdle-related disability, health-related quality of life, Kinesiophobia , global improvement and ASLR-RE angle.

Treatment duration will be eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for the study if they met all the following criteria:

  1. Are between 3 and 12 months postpartum.
  2. Are aged between 20 and 35 years.
  3. Have a body mass index (BMI) < 30 kg/m².
  4. Reported experiencing pelvic girdle pain-defined as pain localized between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints-that either began during pregnancy or persisted after delivery .
  5. Presented with a positive Active Straight Leg Raise (ASLR) test.
  6. Showed positive findings in at least two of the following six pelvic pain provocation tests:

     * Posterior Pelvic Pain Provocation (P4/Thigh Thrust) Test
     * Patrick's (FABER) Test
     * Long Dorsal Sacral Ligament Test
     * Pelvic Compression Test
     * Pelvic Distraction (Separation) Test
     * Sacral Thrust Test

Exclusion Criteria:

* -Patients will be excluded if they have any of the following:

  1. If they were Pregnant
  2. Known causes of pelvic girdle pain, such as fractures and rheumatism
  3. Undergone lumbar or pelvic surgery in the past
  4. Current neurological symptoms and signs in lower extremities such as lumbar radiculopathy and myelopathy
  5. Cancer
  6. Cardiovascular disease
  7. Experience with structured and supervised core or trunk exercise training programs

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
pelvic girdle pain intensity ( pain index ) | Baseline , 8 weeks and 16 weeks
  In this study, pain severity will be measured using the mean of three 11-point NRS questionnaires for least, usual, and current pain over the previous 2 weeks.

SECONDARY OUTCOMES:
pelvic girdle-related disability | Baseline , 8 weeks and 16 weeks
  pelvic girdle-related disability, measured by pelvic girdle questionnaire (PGQ)
Health-related quality of life | Baseline , 8 weeks and 16 weeks
  Health-related quality of life, measured by the Arabic version of European quality of life-Five-Dimension Five-Level Instrument (EQ-5d-5L)
Kinesiophobia | Baseline , 8 weeks and 16 weeks
  Kinesiophobia measured by an Arabic Tampa scale
Global improvement | Baseline , 8 weeks and 16 weeks
  Global improvement measured by global rating of change (GROC) scale
Active straight leg raises repositioning error (ASLR-RE) | Baseline , 8 weeks and 16 weeks
  ASLR-RE angle, measured by Image J